CLINICAL TRIAL: NCT02506530
Title: Contribution of an Endermologie LPG Cellu M6 Treatment in the Treatment Pathway of Patients Suffering From a Breast Cancer Related Lymphoedema, During an Intensive Decongestive Treatment.
Brief Title: Treatment Pathway of Patients Suffering From a Breast Cancer Related Lymphoedema
Acronym: ELOCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Collaborators: LPG SYSTEMS (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC31/14/7425
Record Dates: First submitted 2015-07-16; First posted 2015-07-23 (Estimated); Last update posted 2025-12-05 (Actual); Status verified 2019-08

CONDITIONS: Lymphedema
Keywords: lymphedema; breast cancer
MeSH Terms: conditions — Lymphedema; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- intensive decongestive treatment (IDT) (Active Comparator): Patients will receive an intensive decongestive treatment for 5 days
  Interventions: Procedure: intensive decongestive treatment
- IDT + Cellu M6 (Experimental): Patients will receive an intensive decongestive treatment + Cellu M6 for 5 days
  Interventions: Procedure: intensive decongestive treatment; Device: Cellu M6
- Cellu M6 + bandages (Active Comparator): Patients will receive an bandages + Cellu M6 for 5 days
  Interventions: Device: Cellu M6

INTERVENTIONS:
Procedure: intensive decongestive treatment — intensive decongestive treatment
  Arms: IDT + Cellu M6; intensive decongestive treatment (IDT)
Device: Cellu M6 — Use of Cellu M6
  Arms: Cellu M6 + bandages; IDT + Cellu M6

SUMMARY:
This study will assess the benefit of LPG Cellu M6 in addition of intensive decongestive treatment in reducing secondary lymphoedema in breast cancer.

DETAILED DESCRIPTION:
The main objective of the study is to assess the proportion of successfully treated patients (success rate).

That is to say patients having a reduction of excess arm volume ≥ 30% after 5 days of three types of treatment for secondary lymphoedema :

Group 1: standard intensive decongestive therapy for 5 days (bandages + manual lymphatic drainage).

Group 2: standard intensive decongestive therapy (bandages + manual lymphatic drainage) + Cellu M6 for 5 days Group 3: Bandages + Cellu M6 for 5 days

Symptomatic treatment of lymphoedema reference is intensive decongestive therapy including manual lymphatic drainage, compression of multicomponent bandaging, therapeutic exercise and skin care (HAS 2012 ISL International Society of Lymphology, 2013).

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from a lymphoedema consequence of a breast cancer of grades 2 or 3 (ISL)
* Patients suffering from Lymphoedema for 6 months or more
* Patients with a difference between arms >10%
* Patients who had ever had an axillary node dissection
* Patients hospitalized for intensive standard treatment.

Exclusion Criteria:

* Primary lymphoedema
* Venous insufficiency of the upper members
* severe arterial obstruction
* obliterating arteritis of the upper limbs
* Bilateral lymphoedema
* Breast cancer recurrence
* Another cancer in treatment
* Decompensated heart failure
* Pacemaker
* acute infection
* Deep venous thrombosis
* Skin atrophy of the upper member
* Bullous dermatosis
* Acute dermatitis with epidermitis or dermatitis-hypodermitis
* Infected wound
* Inflammatory scar or consequence of a recent surgery (<1 month)
* Presence of osteosynthesis equipment under the skin with an external part in the upper member to treat
* Hyperalgesia of the shoulder
* Pregnancy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
The proportion of patients successfully treated (reduction of the excessive volume in the arm>30%) | 6 months

SECONDARY OUTCOMES:
Progression of the excessive volume in the arm since hospitalization | 6 months
assess adverse effects | 6 months

OTHER OUTCOMES:
cost effectiveness analysis of treatments | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Julie MALLOIZEL-DELAUNAY, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- MALLOIZEL DELAUNAY Julie, Toulouse, Midi Pyrenees, France

REFERENCES:
- [Result] Malloizel-Delaunay J, Chantalat E, Bongard V, Chaput B, Garmy-Susini B, Yannoutsos A, Vaysse C. Endermology treatment for breast cancer related lymphedema (ELOCS): Protocol for a phase II randomized controlled trial. Eur J Obstet Gynecol Reprod Biol. 2019 Oct;241:35-41. doi: 10.1016/j.ejogrb.2019.07.040. Epub 2019 Aug 7. PMID 31419694
- [Result] Malloizel-Delaunay J, Weyl A, Brusq C, Chaput B, Garmy-Susini B, Bongard V, Vaysse C. New Strategy for Breast Cancer Related Lymphedema Treatment by Endermology: ELOCS Phase II Randomized Controlled Trial. Clin Breast Cancer. 2024 Aug;24(6):533-540. doi: 10.1016/j.clbc.2024.05.009. Epub 2024 May 22. PMID 38853038